CLINICAL TRIAL: NCT02839564
Title: Benefit of Laparoscopic Adhesiolysis
Brief Title: Benefit of Laparoscopic Adhesiolysis in Patients With Chronische Abdominal Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Groene Hart Ziekenhuis (Other)
Collaborators: Erasmus Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Rijnstate Hospital (Other); Maxima Medical Center (Other); Catharina Ziekenhuis Eindhoven (Other); Maasstad Hospital (Other); Isala (Other)
Responsible Party: Principal Investigator, Marijke Molegraaf, Drs, Groene Hart Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 160.613/1997/70
Record Dates: First submitted 2016-07-14; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Pain; Adhesions
Keywords: chronic abdominal pain; laparoscopic adhesiolysis; placebo
MeSH Terms: conditions — Chronic Pain; Tissue Adhesions | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adhesiolysis group (Experimental): Patients underwent laparoscopic adhesiolysis
  Interventions: Procedure: Laparoscopic adhesiolysis
- Placebo group (Placebo Comparator): Patients underwent diagnostic laparoscopy alone
  Interventions: Procedure: Diagnostic laparoscopy

INTERVENTIONS:
Procedure: Laparoscopic adhesiolysis — After diagnostic laparoscopy to confirm adhesions and exclude other pathology laparoscopic adhesiolysis was performed
  Arms: Adhesiolysis group
Procedure: Diagnostic laparoscopy — After diagnostic laparoscopy to confirm adhesions and exclude other pathology treatment was stopped.
  Arms: Placebo group

SUMMARY:
Laparoscopic adhesiolysis as a therapy for chronic pain is still controversial and long term effects are not known. The objective was to to evaluate long term effects of laparoscopic adhesiolysis for treating chronic abdominal pain.

Therefore one hundred patients with abdominal pain attributed to adhesions were randomized to laparoscopic adhesiolysis or a placebo group with laparoscopy alone. Pain relief was assessed after 3, 6 and 12 months and 12-year follow-up.

DETAILED DESCRIPTION:
This multi-center randomized controlled trial, included patients with chronic abdominal pain likely to be caused by adhesions from previous abdominal surgery. Chronic abdominal pain was defined as continues or intermittent abdominal pain of at least six months' duration. After excluding other pathology (see exclusion criteria) included patients underwent a diagnostic laparoscopy to confirm the adhesions and to exclude serious morbidity not visible with other diagnostics. If during laparoscopy adhesions were the only pathology present, patients were randomly assigned either to laparoscopic adhesiolysis or no treatment. For the randomization and surgical procedures the investigators refer to the original article. Patients were unaware of their treatment assignment and the outcome assessment was blinded. Abdominal pain and quality of life (QOL) were assessed pre-operatively and at 3, 6 and 12 months of follow-using a visual analog scale (VAS), verbal rating pain change score (VRCS) and the short form 36 (SF-36). After twelve months randomization was disclosed and placebo group patients with persisting abdominal pain could request laparoscopic adhesiolysis. After twelve year follow-up pain, QOL, medical history and analgesic intake were analyzed to assess the long term effects of laparoscopic adhesiolysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above with chronic abdominal pain that was likely to be caused by adhesions due to previous abdominal surgery were recruited. Before attributing abdominal pain to the existence of adhesions all patients had an extensional diagnostic work-up to exclude other pathology.

Exclusion Criteria:

* Current treatment by psychologist or psychiatrist
* Use of laxatives, sedatives, morphine, antipsychotics, antidepressants, or drugs that stimulate the central nervous system
* Abnormal outcome of standardized non-invasive diagnostics:

  * Biochemical investigation
  * Lactose tolerance tests or H2 respiration test
  * Feces analysis of worms and worm eggs
  * Ultrasound or CT scan of the abdomen
  * Radiographic studies of small and large bowel (or colonoscopy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1997-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Short term pain relief | 12 months
  Pain relief was assessed using a verbal rating pain change score (VRCS)
Long term pain relief | 12 year
  Pain relief was assessed using a verbal rating pain change score (VRCS)

SECONDARY OUTCOMES:
Quality of life | 12 months and 12 year
  QOL was assessed using the Short Form 36
Complications of treatment | 12 year
Analgesic intake | 12 months and 12 year
additional surgery because of persisting abdominal pain | 12 months and 12 year
  patient questionnaire, patients medical record
rate of consulting medical doctors | 12 months and 12 year

CONTACTS AND LOCATIONS:
Overall Officials: Dingeman Swank, Dr, Principal Investigator — Groene Hart Ziekenhuis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Swank DJ, Swank-Bordewijk SC, Hop WC, van Erp WF, Janssen IM, Bonjer HJ, Jeekel J. Laparoscopic adhesiolysis in patients with chronic abdominal pain: a blinded randomised controlled multi-centre trial. Lancet. 2003 Apr 12;361(9365):1247-51. doi: 10.1016/s0140-6736(03)12979-0. PMID 12699951
- Available data/document: Study Protocol — http://gmail.com — Study data can be requested by mailing to mjmolegraaf@gmail.com